CLINICAL TRIAL: NCT02403492
Title: Treatment of Obstructive Sleep Apnea in Children: An Opportunity for Cardiovascular Risk Modification
Acronym: TREAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Indra Narang, Director, Sleep Medicine, Staff Pulmonologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1000026523
Record Dates: First submitted 2014-12-22; First posted 2015-03-31 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Obesity; Obstructive Sleep Apnea; Sleep Disorders; Cardiovascular Disease
Keywords: Children; Obesity; Cardiovascular; Sleep; Apnea; Obstructive
MeSH Terms: conditions — Obesity; Sleep Apnea, Obstructive; Sleep Wake Disorders; Cardiovascular Diseases; Apnea | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Observational (No OSAS) (No Intervention): Comprised of obese children are not found to have obstructive sleep apnea and do not require cPAP
- Experimental - cPAP, Continuation (Experimental): Comprised of those obese children who are diagnosed with obstructive sleep apnea, requiring cPAP, who continue using cPAP during the 2 week RCT
  Interventions: Device: cPAP; Device: cPAP, Continuation
- Experimental - cPAP Discontinuation (Experimental): Comprised of those obese children who are diagnosed with obstructive sleep apnea, requiring cPAP, who discontinue using cPAP during the 2 week RCT
  Interventions: Device: cPAP; Device: cPAP, Discontinuation

INTERVENTIONS:
Device: cPAP — All participants diagnosed with obstructive sleep apnea will be required to use cPAP for 6 months prior to the RCT component of this trial
  Other Names: continuous Positive Airway Pressure
  Arms: Experimental - cPAP Discontinuation; Experimental - cPAP, Continuation
Device: cPAP, Continuation — Participants will be randomized to continue cPAP for a 2 week period
  Arms: Experimental - cPAP, Continuation
Device: cPAP, Discontinuation — Participants will be randomized to discontinue cPAP for a 2 week period
  Arms: Experimental - cPAP Discontinuation

SUMMARY:
Heart disease is a major cause of ill-health and death in adults. The risk factors for heart disease, if present in children, carry over into adult life. Childhood obesity has reached epidemic proportions in Canada and is associated with many heart disease risk factors such as high blood pressure. Another complication of obesity is obstructive sleep apnea. Sleep apnea is marked by snoring at night, pauses in breathing and low oxygen levels and occurs in up to 60% of obese children, but it is diagnosed in less than 20% of obese children. Importantly, sleep apnea in children, like obesity, is linked with high blood pressure and heart disease. Thus, children with sleep apnea who are obese are likely to have an increased risk for high blood pressure and heart disease. Currently, there is little knowledge of the extent of heart disease in obese children with sleep apnea.

The best treatment for both obesity and sleep apnea is weight loss. Weight loss strategies are generally not very successful and since 75% of obese children will become obese adults, urgent treatments are needed to reduce heart disease in the long-term. Treating sleep apnea in obese children may be one of the ways to reduce heart disease. Sleep apnea can be treated with continuous positive airway pressure (CPAP), which involves wearing a mask attached to a breathing machine while asleep. It is unknown how effective CPAP is in reducing heart disease in obese children.

The investigators will recruit children with sleep apnea who are obese and test for heart disease risk. The investigators will then treat these children with CPAP. After 6 months of CPAP, the investigators will repeat the tests to determine if CPAP lowers the risk for heart disease. At the end of the 6 months, those receiving CPAP will be randomized to either continue CPAP or discontinue CPAP for a 2 week period. At the end of the 2 week period the participants will repeat the tests again to determine the magnitude of the effect of CPAP.

The investigators expect that CPAP treatment for sleep apnea in obese children will reduce blood pressure and lower heart disease. These results will increase awareness of the dangers of sleep apnea in obese children, which will facilitate early diagnosis and treatment, ultimately reducing heart disease long-term.

DETAILED DESCRIPTION:
Statement of the Problem: In Canada, child and adolescent obesity, defined as a body mass index (BMI) of >95th percentile for age and gender1 represents one of the most common conditions effecting children in Canada with an obesity rate of 10% in 12-17 year old children, which currently equates to approximately half a million obese children in Canada. Obesity is not only complicated by cardiovascular and metabolic dysfunction, such as left ventricular modeling, hypertension, glucose intolerance and dyslipidaemia, it is also associated with obstructive sleep apnea syndrome (OSAS), occurring in up to 60% of obese children.

OSAS is characterized by snoring, recurrent partial (hypopneas) or complete obstruction (apneas) of the upper airway, frequently associated with intermittent oxyhaemoglobin desaturations, sleep disruption and fragmentation. The gold standard test for diagnosing obstructive sleep apnea is a polysomnogram (PSG). Specifically, OSAS affects 1-4% of healthy children who are typically 2-8 years of age6, coinciding with adenotonsillar hypertrophy, the commonest cause of OSAS in children. Usual treatment for OSAS in children with adenotonsillar hypertrophy is an adenotonsillectomy (AT). However, there is clear evidence that not only is there a high prevalence of obstructive sleep apnea in obese children, but further, the AT is not successful for resolution of OSAS. This is, in part due to the fact that adenotonsillar hypertrophy is not the single most significant risk factor for OSAS in the obese population.

The factors implicated in the pathophysiology of OSAS in obese children include soft tissues restricting the upper airway size such as fat pads in the soft palate, lateral pharyngeal wall and at the base of the tongue. However, despite the anatomic evidence predisposing obese children to OSAS there are also alterations in functional mechanisms that lead to increased airway collapsibility predisposing these children to OSAS. Specifically, obesity is associated with significant alterations in body composition that could affect chest wall mechanics by weighting the chest wall and reducing lung compliance. Functional residual capacity is diminished to abdominal visceral fat impinging on the chest cavity. Such a reduction in functional residual capacity and compliance increases the risk for sleep disordered breathing by mechanisms of hypoventilation, atelectasis and ventilation perfusion mismatch all increasing the work of breathing and fatigue. Moreover, hypoventilation in itself may reduce upper airway motor tone. Further, ventilator responses may be altered as studies focusing on obese adults have shown that morbidly obese subjects are more susceptible to decreased ventilatory responses to both hypoxia and hypercapnia.

Given this understanding that adenotonsillectomy is not curative in obese children with obstructive sleep apnea, weight loss would be considered the treatment of choice. However, obesity intervention programs have not been wholly successful in BMI reduction in children although in overweight adults, magnitude of weight loss was related to an improvement in OSAS. Thus, the delivery of positive airway pressure (PAP) either continuous positive airway pressure (CPAP) or bilevel positive airway pressure (BiPAP) is increasingly used as the first line of treatment for OSAS in obese children, although usually in conjunction with weight loss strategies.

Although the benefits of PAP are well established in adults, there is a paucity of available paediatric data.

As previously mentioned, obesity is a risk factor for cardiovascular and metabolic dysfunction; however, OSAS independent of obesity is further associated with cardiac remodeling and cardiovascular metabolic dysfunction. Specifically, if untreated, obstructive sleep apnea in children may lead to excessive daytime sleepiness, poor school performance, hypertension, changes in left ventricular mass and geometry, endothelial cell dysfunction, arterial stiffness, autonomic dysfunction inflammation, and the Metabolic Syndrome (MetS). Thus, OSAS in the context of obesity may independently or synergistically magnify the risk of an already compromised cardiometabolic regulation.

Several metrics will be utilized. Physical activity levels will be measured utilizing Habitual Activity Questionnaires. Insulin resistance will be measured using Fasting Glucose and Fasting Insulin Levels. Cardiovascular markers will include 24 hour blood pressure and cardiograms - left ventricular mass index. C Reactive Protein (CRP) will be utilized as the marker of inflammation.

The mechanisms linking both OSAS and obesity to cardiometabolic dysfunction is believed to be due to activity of the sympathetic nervous system (SNS) and effects of oxidative stress, exacerbating proinflammatory states. Chronic, awake sympathoactivation may promote vascular remodeling and can induce significant cardiovascular morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Obesity, BMI > 95th centile for age and gender
* 10-18 years of age
* Informed consent and the ability to perform the tests
* Moderate to sever OSAS (will be eligible for inclusion in the treatment group for this study)

Exclusion Criteria:

* Use of anti-hypertensive medication
* Medications known to alter glucose and insulin regulation
* Significant central sleep apnea
* Currently unwell or recent viral/bacterial infection in the previous 4 weeks
* Currently hospitalized
* Known underlying neuromuscular disorder, congenital heart disease, diagnosed ventricular disorder
* Syndrome's e.g. Down (high prevalence of OSAS independent of obesity)
* Pregnancy
* Gastric bypass surgery
* Unable to have a PSG perfumed for whatever reason

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Actual)
Dates: Start 2013-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
To assess changes in cardiovascular markers pre and post PAP therapy | Baseline, 6 Months
  To assess the efficacy of PAP therapy for OSAS in obese children on left ventricular mass index.

SECONDARY OUTCOMES:
To evaluate changes in health-related quality of life prior to and post treatment with PAP therapy for OSAS. | Baseline, 6 Months
To assess the efficacy of PAP therapy for OSAS in obese children on heart rate variability. | Baseline, 6 Months
To determine changes in blood pressure in obese children with OSAS prior to and post treatment with PAP therapy. | Baseline, 6 Months
To assess the efficacy of PAP therapy for OSAS on changes in insulin resistance in obese children. | Baseline, 6 Months
To assess the efficacy of PAP therapy for OSAS in obese children on changes in vascular structure using pulse wave velocity. | Baseline, 6 Months
To assess changes in C Reactive Protein (CRP) markers pre and post PAP therapy in obese children with OSAS. | Baseline, 6 Months

OTHER OUTCOMES:
To assess the efficacy of PAP therapy for OSAS in obese children on changes in physical activity levels. | Baseline, 6 Months
To assess the efficacy of PAP therapy for OSAS in obese children on changes in sleep duration. | Baseline, 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Indra Narang, MD, FRCPCH, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada